CLINICAL TRIAL: NCT05619029
Title: Retrospective, Observer-blinded, Pivotal Study to Evaluate the Effectiveness of the Investigational Device (Lunit INSIGHT CXR) in Detection of Abnormal Findings on Chest Radiographs
Brief Title: Study to Evaluate the Effectiveness of the Device in Detection of Abnormal Findings on X-ray
Status: Completed | Type: Observational
Sponsor: Lunit Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LUN_CXR_CA_222
Record Dates: First submitted 2022-11-02; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive: chest radiographs with the specific target radiologic findings (Atelectasis, Calcification, Cardiomegaly, Consolidation, Fibrosis, Mediastinal Widening, Nodule/Mass, Pleural Effusion, Pneumoperitoneum, Pneumothorax)
  Interventions: Radiation: X-ray
- Negative: chest radiographs with no target radiologic findings
  Interventions: Radiation: X-ray

INTERVENTIONS:
Radiation: X-ray — Chest radiographs

SUMMARY:
This study aims to evaluate the effectiveness of the investigational device (Lunit INSIGHT CXR) in the detection of chest abnormalities.

DETAILED DESCRIPTION:
In the study, the standalone performance of Lunit INSIGHT CXR was primarily assessed by comparing the analysis results from the investigational device and reference standards in the detection of 10 abnormal radiologic findings - atelectasis, calcification, cardiomegaly, consolidation, fibrosis, mediastinal widening, nodule/mass, pleural effusion, pneumoperitoneum, and pneumothorax.

In addition, to investigate the effect of Lunit INSIGHT CXR assistance on the interpreting physician's interpreting performance, a multi-reader, multi-case (MRMC) study was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiographs of aged 14 years or older
* Conventional PA or AP chest radiographs
* Chest radiographs with confirmed radiology reports

Exclusion Criteria:

* Chest radiographs taken in postures other than PA and AP e.g.) decubitus, oblique, lordotic, or lateral view
* Invert-grayscale chest radiographs
* Image quality not suitable for interpretation due to incorrect patient positioning, inadequate image collimation, severely damaged lung presence of external materials such as jewelry

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The secondary hospital patients
Sampling Method: Probability Sample
Enrollment: 1111 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (ROC AUC) of the investigational device in detection of overall target radiologic findings | Through study completion, an average of 6 months
  To evaluate the effectiveness of the investigational device (Lunit INSIGHT CXR) in the detection of chest abnormalities, Area Under the Receiver Operating Characteristic Curve (ROC AUC) of the investigational device in detection of overall target radiologic findings (detection of any abnormal findings among ten target radiologic findings) will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No